CLINICAL TRIAL: NCT01610323
Title: Fitness Improvement in Obese, Pregnant Women: an Intervention Trial (InterGOFIT)
Brief Title: Fitness Improvement in Obese, Pregnant Women: an Intervention Trial
Acronym: InterGOFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Foundation of the Stars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SC11-05-021-21
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Pregnancy; Obesity; Physical Activity
Keywords: Pregnancy; Obesity; Physical activity; Cardiorespiratory fitness; Muscular Fitness; Weight gain; Fetal growth
MeSH Terms: conditions — Obesity; Motor Activity; Weight Gain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental): Exercise intervention
  Interventions: Other: Exercise intervention
- Control group (Other): Standard care
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Exercise intervention — Exercise group: 12 weeks of moderate intensity physical training under individual supervision in a specialised conditioning center, with a goal of 3 1h-sessions/week (from 16 wks to 28 wks of gestation). Including aerobic and muscular training.
  Other Names: Physical activity intervention
  Arms: Exercise group
Other: Standard Care
  Arms: Control group

SUMMARY:
In pregnancy, the adoption or pursuit of a sedentary lifestyle contributes to the development of co-morbid conditions such as hypertension, maternal and childhood obesity, gestational diabetes, pre-eclampsia, cesarean section and delivery of large-for-gestational-age infants (LGA).

The aim of this study is to test the hypothesis that obese, pregnant women following a supervised moderate intensity physical conditioning program during the 2nd trimester of pregnancy will maintain a higher level of physical activity up to the end of pregnancy, as compared to women in the control group. We will also conduct a pilot study on the feasibility to examine the effects of the intervention on maternal fitness and neonatal anthropometry.

DETAILED DESCRIPTION:
Looking at the multiple needs of pregnant women with obesity, physical conditioning may offer a great opportunity to improve fitness and to decrease cardio-metabolic disturbances, to prevent excessive weight gain, to improve general health status, and to reduce health care utilization. Furthermore, beneficial effects of fitness on adverse maternal health outcomes related to obesity might decrease the development of long-term obesity and metabolic repercussions in the offspring.

The Society of Obstetricians and Gynaecologists of Canada (SOGC) recommends that all women without contraindication be encouraged to participate in aerobic and strength-conditioning exercises as part of a healthy lifestyle during pregnancy. Despite these recommendations, obese women are inactive during pregnancy and are currently still at high risk of poor physical fitness.

Thus, although exercise clearly improves maternal health status and thus potentially prevents adverse perinatal outcomes, obese pregnant women poorly adhere to experts' recommendations about the need for exercise during pregnancy. Therefore, this situation justifies the need to develop adapted strategies aimed at increasing the implementation of guideline recommendations in this population.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 18 years or older
* single pregnancy
* delivery at Centre Hospitalier Universitaire de Québec
* pre-pregnancy BMI ≥30 kg/m2

Exclusion Criteria:

* multiple pregnancy
* diabetes or chronic hypertension prior to pregnancy
* uncontrolled thyroid problems
* exercise contraindications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Weekly time spent at physical activity of moderate intensity and above | At 36 weeks of gestation
  Accelerometry data (minutes per week spent over selected cutpoints)

SECONDARY OUTCOMES:
Gestational weight gain | At 36 weeks of gestation
  Weight in kg at 36 weeks - weight in kg at 14 weeks
Muscular fitness | At 28 wks of gestation
  Endurance and strength of lower and upper limbs as assessed by an isokinetic dynamometer.
Cardiorespiratory fitness | At 28 weeks of gestation
  O2 consumption (ml*kg-1*min-1) at the anaerobic threshold.
Energy Expenditure | At 36 weeks of gestation
  According to the Pregnancy Physical Activity Questionnaire (PPAQ)
Neonatal anthropometry | At delivery
  Birth weight, length and skinfolds
Fetal growth | At 28 weeks of gestation
  Ultrasound and doppler

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Marc, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Québec (CHUQ)
Locations (1):
- Centre Hospitalier Universitaire de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bisson M, Almeras N, Dufresne SS, Robitaille J, Rheaume C, Bujold E, Frenette J, Tremblay A, Marc I. A 12-Week Exercise Program for Pregnant Women with Obesity to Improve Physical Activity Levels: An Open Randomised Preliminary Study. PLoS One. 2015 Sep 16;10(9):e0137742. doi: 10.1371/journal.pone.0137742. eCollection 2015. PMID 26375471